CLINICAL TRIAL: NCT01178580
Title: Procoagulant Activity in Patients With Community Acquired Pneumonia, Pleural Effusion and Empyema
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10-138-10.CTIL
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Pneumonia; Pleural Effusion; Empyema
Keywords: fibrinolytic activity; Community acquired pneumonia (CAP); Pleural effusion
MeSH Terms: conditions — Pneumonia; Pleural Effusion; Empyema; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Community acquired pneumonia (CAP) is still one of the most important causes of morbidity in adults. (1) In severe cases, parapneumonic effusions or empyema may develop. In these patients, a transitional fibrin neomatrix constitutes part of the acute inflammatory response as seen in sepsis.

The aim is to study the fibrinolytic activity in patients with CAP alone versus CAP with parapneumonic effusions with and without empyema.

DETAILED DESCRIPTION:
Community acquired pneumonia (CAP) is still one of the most important causes of morbidity in adults. (1) In severe cases, parapneumonic effusions or empyema may develop. In these patients, a transitional fibrin neomatrix constitutes part of the acute inflammatory response as seen in sepsis. (2) The increased vascular permeability, mediated by several cytokines, such as IL-1, IL-6, IL-8, tumor necrosis factor (TNF), and platelet activator factor, allows migration of inflammatory cells, an increased fluid accumulation and bacterial invasion into pleural space. (3) At this stage, activation of the coagulation cascade leads to procoagulant activity and decreased fibrinolysis with deposition of fibrin in the pleural space. The activation of the fibrinolytic system produce the D-dimer and follow by increased other procoagulant markers like thrombin anti thrombin, fragment 1.2 (4-5) Several studies showed that the plasma D-dimer levels were increased even in community-acquired pneumonia patients. Moreover, others reported that Serum levels of AT-III, D-D and CRP at admission appear to be useful biomarkers for assessing the severity of CAP. However, no data exists about the fibrinolytic profile in patients with CAP alone in compare to CAP with parapneumonic effusion with and without empyema.

Aim:

To study the fibrinolytic activity in patients with CAP alone versus CAP with parapneumonic effusions with and without empyema.

ELIGIBILITY:
Inclusion Criteria:

* All patients that will be admitted with CAP to the pulmonary department in Meir Medical Center and have no exclusion criteria will be included in the study.

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with anticoagulant treatment, primary coagulopathy, nephrotic syndrome, surgery, other infection in the month preceding the study, an abnormal liver or renal function test(s), a history of deep vein thrombosis in the last year or patients with acute coronary syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients that will be admitted with CAP to the pulmonary department in Meir Medical Center and have no exclusion criteria will be included in the study
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shitrit, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Pulmonary department, Meir Medical Center, Kfar Saba, Israel, Israel